CLINICAL TRIAL: NCT01525264
Title: Korean Immigrants & Mammography-Culture-Specific Health Intervention (KIM-CHI)
Brief Title: Breast Cancer Screening Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 10-000204; Kim-CHi (Other Grant/Funding Number: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2011-12-26; First posted 2012-02-02 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culturally Relavent Education (Experimental): Education about improving diet using a DVD with Korean role models and native Korean language.
  Interventions: Behavioral: KIM-CHI
- Healthy Wife Intervention (Active Comparator): Intervention group of couples who received education about importance of a Healthy Diet. It was an attention control group
  Interventions: Behavioral: Healthy Wife Control Group

INTERVENTIONS:
Behavioral: KIM-CHI — The intervention is based on cultural characteristics and context and focuses on changing (1) beliefs about breast cancer and screening, (2) knowledge of breast cancer and screening, (3) self-efficacy of confidence in one's ability to complete all the steps necessary for obtaining a mammogram including requesting a referral for mammogram from a physician. The KIM-CHI program also incorporates strategies for enhancing spousal support (perceived support received from husband). To standardize delivery of culture-relevant health behavior change information related to breast cancer screening to groups of women and their husbands separately, the KIM-CHI program uses a DVD with Korean role models, native Korean language, and male physician authentication as well as inclusion of spouses.
  Other Names: Culturally relavent intervention
  Arms: Culturally Relavent Education
Behavioral: Healthy Wife Control Group — Intervention group of couples who received education about importance of Healthy diet
  Other Names: Healthy Diet
  Arms: Healthy Wife Intervention

SUMMARY:
Breast cancer is the most commonly occurring cancer and most common cause of cancer mortality among Korean American (KA) women, but mammography utilization among KA women remains suboptimal. Most breast cancer screening studies with KA women have been descriptive and correlational. Therefore, in this 4-year project, the effects of Korean Immigrants & Mammography-Culture-Specific Health Intervention (KIM-CHI) on adherence to recommended breast cancer screening protocols were tested. The specific aims are to: (1) compare the group receiving KIM-CHI with an attention control group on mammogram attainment outcomes including number of mammograms obtained (0, 1, or 2) and if obtained, length of time to obtain the first mammogram, at 15 months using survival analysis; (2) compare the two groups on the mediating variables of health beliefs, knowledge, self-efficacy, and spousal support at 2 weeks, 6 months, and 15 months using repeated measures multivariate analysis of variance; and (3) identify the mediating effects of health beliefs, knowledge, self-efficacy, and spousal support at 2 weeks on mammogram attainment outcomes at 15 months, using structural equation modeling. Data on mammography attainment and the mediating variables were collected at baseline and at 2-weeks, and 6- and 15-months post-baseline.

DETAILED DESCRIPTION:
In this two-group cluster randomized, longitudinal, controlled design, the KIM-CHI and control activities were delivered immediately after baseline data collection at 50 KA religious organizations. Participants in the attention control group followed the same study procedures as participants in the KIM-CHI group, except for the content of the educational films. The baseline and longitudinal data were collected from August 2008 to September 2010 in Cook County, Illinois.

The KIM-CHI group slogan was "Healthy Family, Healthy Wife," and the control group slogan was "Healthy Family, Healthy Diet," emphasizing the importance of the husband's support in promoting family health by improving breast cancer screening or diet in the KIM-CHI and attention control groups, respectively.

The KIM-CHI program consisted of (1) showing a project team-designed 30-minute Korean language film (in DVD format) on breast cancer screening to change health beliefs; (2) holding a brief group discussion session immediately after the film showing; and (3) requiring each couple to complete a discussion activity together at home to enhance spousal support for the women.

A total of 516 women were assessed for eligibility for this study from August 2008 to June 2009. 428 KA women were recruited at baseline. The response rates for returning homework activity in intervention and control groups were 98.1% (207/211) and 98.6% (214/217), respectively.

All the variables reported are from KA women, but socio-demographic variables are from both KA women and their husbands. Mammography uptake was measured by self-report at 6- months and 15-months post-baseline, based on the ACS guideline recommending that women 40 and older receive a mammogram every year. Predictor variables measured were age, education, employment, and level of acculturation. Level of acculturation was measured by the Suinn-Lew Asian Self-Identity Acculturation Scale (SL-ASIA). The SL-ASIA was modified slightly by deleting one item about generation because it was not relevant for first-generation KAs. The words "Asian" and "Oriental" in the original instrument were also changed to "Korean." Scoring for the revised SL-ASIA was the same as the original SL-ASIA, using a 5-point Likert scale with a final score ranging from 1.00 (low acculturation) to 5.00 (high acculturation). Questions on health care resources and utilization, health insurance status, usual source of care (a regular place or doctor to visit), and physical examinations in the past 2 years without sickness or for health problems were measured. Family history of breast cancer and history of mammography (when the last mammogram was, if they ever had one) were also measured.

After Human Subjects Review Approval was obtained, invitation letters were mailed to all 210 religious organizations listed in the Korean language Chicago Korean Business Directory 2006. One hundred KA organizations were contacted to request participation in the study and 110 KA religious organizations were treated as "unable to reach." Of those 100 contacted organizations, 32 were ineligible (e.g., they were younger KAs, students, multi-ethnics, or disabled persons). Eighteen of the remaining 68 eligible organizations (26.5%) refused to participate. The 50 organizations were randomly assigned to either the KIM-CHI or attention control group. After random assignment, the characteristics of religious organizations (location and size) were not statistically significantly different between the two groups.

A total of 428 couples participated in this study at baseline; 211 wife-husband dyads from 26 KIM-CHI organizations and 217 wife-husband dyads from 24 attention control organizations. KA women and their husbands who were interested in participating in our study signed two copies of an informed consent form. Next, each completed a self-administered baseline questionnaire which took 30-45 minutes. Then they received the KIM-CHI or control education.

Six- and 15-month post-baseline data were collected via phone by telephone surveyors who were blind to the study group assignment. At 6-months, 414 women participated in the telephone survey in Korean, with 3.3% lost to follow-up. At 15-months post-baseline, 395 women participated in the telephone survey, with 7.7% lost to follow-up, for the entire study period. The reasons for lost to follow-up were death, refused to participate, or unable to contract. KA women included at the 15 months' data collection (n = 395) and those who dropped out (n = 33) did not differ in demographic or other major variables in this study.

ELIGIBILITY:
Inclusion Criteria:

* For women, criteria for inclusion in the study are

  1. 40 years of age or older
  2. born in Korea but presently living in the U.S.
  3. able to speak and read Korean
  4. married to a KA man who meets inclusion criteria (2) and (3).

Exclusion Criteria:

* Women who have had a mammogram within the past 1 year or have been diagnosed with breast cancer were excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mammography uptake at 15 months | 6- and 15-months post-baseline
  Non of the participants at baseline had a mammogram within the previous 1 year. The primary outcome was measured by self-report about how many times and when (month and year) mammograms were obtained by women in the study, with follow-up validation by the mammography facility for each woman who reports having had a mammogram in the past 15 months at Time 3. The number of mammograms (o, 1, or 2) and length of time to mammogram were calculated.

SECONDARY OUTCOMES:
Health beliefs | 6- and 15-months post-baseline
  health beliefs (perceived seriousness, susceptibility, benefits, barriers, knowledge, self-efficacy about breast cancer and screening) were measured by using Likert-type scale, ranging from strongly disagree = 1 to strongly agree = 5.
Spousal Support | 6- and 15-months post-baseline
  Women's perceived spousal support received from husbands and husbands' perceived spousal support provided to their wives were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Eunice E Lee, PhD, Principal Investigator — UCLA School of Nursing